CLINICAL TRIAL: NCT02329457
Title: Efficacy and Safety of a Novel Intradermal Live-attenuated Varicella Zoster Vaccine in Hematopoietic Stem Cell Transplantation Donors: a Randomized Double Blind Placebo-controlled Trial
Brief Title: VZV Vaccine for Hematopoietic Stem Cell Transplantation
Acronym: VZIDST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HKU 11-174
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Varicella Zoster Infection
Keywords: double-blind, randomized, intradermal, VZVv, HSCT
MeSH Terms: conditions — Varicella Zoster Virus Infection | interventions — Herpes Zoster Vaccine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ID varicella zoster vaccine (VZVv) group (Experimental): intradermal 0.65 mL Zostavax
  Interventions: Biological: Zostavax
- SC VZVv group (Active Comparator): subcutaneous 0.65 mL Zostavax
  Interventions: Biological: Zostavax
- ID NS Group (Placebo Comparator): intradermal 0.65 mL normal saline
  Interventions: Biological: Normal Saline
- SC NS Group (Placebo Comparator): subcutaneous 0.65 mL normal saline
  Interventions: Biological: Normal Saline

INTERVENTIONS:
Biological: Zostavax — varicella zoster vaccine
  Arms: ID varicella zoster vaccine (VZVv) group; SC VZVv group
Biological: Normal Saline — normal saline placebo vaccine
  Arms: ID NS Group; SC NS Group

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) is well-established therapy for patients with malignant hematological diseases. Varicella zoster virus (VZV) reactivation, clinically manifested as herpes zoster (HZ), is a major complication that affects up to 50% of patients. Most patients will require hospitalization. Despite treatment with high dose acyclovir, patients may develop severe complications including the disabling postherpetic neuralgia, corneal ulceration, viral dissemination and secondary bacterial infection. The median onset of infection is the fifth month following transplantation, with 91% of cases occurring within the first year. Direct vaccination of transplants recipients with subcutaneous live-attenuated VZVv before transplantation and up to one year after transplantation is contraindicated. A small prospective non-randomized study has demonstrated that subcutaneous vaccination for donors before HSCT may offer some protection against VZV reactivation in the recipients. Recently, dose-sparing influenza vaccine delivered via a novel intradermal microneedle has been shown to elicit a good immunogenic response in both healthy and elderly subjects. We sought to assess the efficacy and safety of the novel intradermal live-attenuated VZVv in sibling donors undergoing HSCT.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is well-established therapy for patients with malignant hematological diseases. Varicella zoster virus (VZV) reactivation, clinically manifested as herpes zoster (HZ), is a major complication that affects up to 50% of patients. Most patients will require hospitalization. Despite treatment with high dose acyclovir, patients may develop severe complications including the disabling postherpetic neuralgia, corneal ulceration, viral dissemination and secondary bacterial infection. The median onset of infection is the fifth month following transplantation, with 91% of cases occurring within the first year. Direct vaccination of transplants recipients with subcutaneous live-attenuated VZVv before transplantation and up to one year after transplantation is contraindicated. A small prospective non-randomized study has demonstrated that subcutaneous vaccination for donors before HSCT may offer some protection against VZV reactivation in the recipients. Recently, dose-sparing influenza vaccine delivered via a novel intradermal microneedle has been shown to elicit a good immunogenic response in both healthy and elderly subjects. We sought to assess the efficacy and safety of the novel intradermal live-attenuated VZVv in sibling donors undergoing HSCT.

We plan to enroll 160 pairs of adult donors and patients who undergo allogeneic HLA matched sibling HSCT in this prospective randomized double-blind placebo-controlled trial over a period of 3 years. Enrolled donors and patients will be randomized into 4 groups: Group 1: intradermal full dose live-attenuated VZVv; Group 2: subcutaneous full dose live-attenuated VZVv; Group 3: intradermal 0.9% normal saline as control; Group 4: subcutaneous 0.9% normal saline as the second control

All vaccines will be given to the donors within 28 days before HSCT. All intradermal vaccines will be given via a microneedle syringe. Both the investigators and participants will be blinded to the randomization process. The primary end point is the occurrence of HZ in the patients within 12 months of transplantation. The secondary end points are the safety and immunological response in the patients and donors.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing allogeneic hemopoietic stem cell transplant
* HLA identical sibling donors
* participants willing to provide written informed consents

Exclusion Criteria:

* history of zoster in the 12 months prior to transplantation
* exposure to VZV within 4 weeks of transplantation
* neomycin sensitivity
* sensitivity to any components of the zoster vaccine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Herpes Zoster Reactivation | 12 months post transplantation
  Incidence of herpes zoster in stem-cell transplant recipients

SECONDARY OUTCOMES:
Immunological response in recipients | 30, 90, 180 and 360 days post transplantation
  Geometric mean concentration of anti-VZV antibody (IU/mL)
Immunological response in donors | 30, 90, 180 and 360 days post transplantation
  Geometric mean concentration of anti-VZV antibody (IU/mL)
Adverse reaction | 21 days after vaccination
  Rate of adverse reaction in donors after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- Ivan Hung, Hong Kong, Hong Kong

REFERENCES:
- [Result] Hata A, Asanuma H, Rinki M, Sharp M, Wong RM, Blume K, Arvin AM. Use of an inactivated varicella vaccine in recipients of hematopoietic-cell transplants. N Engl J Med. 2002 Jul 4;347(1):26-34. doi: 10.1056/NEJMoa013441. PMID 12097537
- [Result] Leung AY, Chow HC, Kwok JS, Lui CK, Cheng VC, Yuen KY, Lie AK, Liang R. Safety of vaccinating sibling donors with live-attenuated varicella zoster vaccine before hematopoietic stem cell transplantation. Bone Marrow Transplant. 2007 Jun;39(11):661-5. doi: 10.1038/sj.bmt.1705673. Epub 2007 Apr 9. PMID 17417658